CLINICAL TRIAL: NCT03494582
Title: Trans Vaginal Sacrospinous Hysteropexy Versus Abdominal Sacral Hysteropexy for the Management of Uterine Prolapse
Brief Title: Abdominal Versus Vaginal Hysteropexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hamdy Ahmed Saaid, Fellow of OBS/GYN, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVVCP
Record Dates: First submitted 2018-03-29; First posted 2018-04-11 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Uterine Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral Hysteropexy (Experimental): Abdominal approach for uterine suspension
  Interventions: Procedure: Sacral Hysteropexy
- sacrospinous Hysteropexy (Experimental): Transvaginal approach for uterine suspension
  Interventions: Procedure: sacrospinous Hysteropexy

INTERVENTIONS:
Procedure: Sacral Hysteropexy — Abdominal approach for uterine suspension
  Arms: Sacral Hysteropexy
Procedure: sacrospinous Hysteropexy — Transvaginal approach for uterine suspension
  Arms: sacrospinous Hysteropexy

SUMMARY:
This study will compare the vaginal versus the abdominal approach for the management of uterine prolapse

DETAILED DESCRIPTION:
this study compares The unilateral sacrospinous hysteropexy with prolene sutures versus the abdominal sacral hysteropexy using Mersilene suture for the management of uterine prolapse

ELIGIBILITY:
Inclusion Criteria:

* Uterine Prolapse

Exclusion Criteria:

* Previous prolapse surgery Hereditary Connective tissue disorders

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pelvic organ prolapse quantification system | 3 month
  compare Pelvic organ prolapse quantification system between groups

SECONDARY OUTCOMES:
Perioperative data | 1 day
  operative time
operative details | 1 day
  blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy HA Ahmed, MD, Principal Investigator — Ain Shams University
Locations (1):
- Urogynecology Unit, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided